CLINICAL TRIAL: NCT00689416
Title: Exploratory Study of New Imaging Biomarkers for Measurement of Carotid Plaque Inflammation
Brief Title: Effects of Crestor on Inflammation of Atherosclerotic Plaques
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Björn Carlsson, MD, PhD, Medical Science Director, Discovery Medicine CDT, AstraZeneca R&D Mölndal, Sweden
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D4411M00010
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2009-06

CONDITIONS: Atherosclerosis; Inflammatory Activity in Carotid Arteries
Keywords: imaging biomarkers; MRI; FDG-PET/CT scanning; Crestor
MeSH Terms: conditions — Atherosclerosis | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: rosuvastatin
- 2 (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: rosuvastatin — 40 mg, tablet, once daily for 3 months.
  Other Names: Crestor
  Arms: 1
Drug: placebo — 40 mg, tablet, once daily for 3 months
  Arms: 2

SUMMARY:
The primary aim of this study is to investigate the effect of 40 mg dose of rosuvastatin on carotid plaque inflammation measured with MRI and PET scanning, to evaluate whether these techniques are promising for future proof of principle studies. A number of patients will receive placebo as a control.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a non-calcified plaque of at least 2 mm over an at least 6 mm length on first MR scan with an uptake of contrast agent on the dynamic MRI scan
* Signed written Informed Consent.
* Healthy men 18 - 70 years, women 60 - 70

Exclusion Criteria:

* Use of a statin within six months before randomization.
* Use of lipid altering medication other than statins within the last six months.
* Clinical evidence of metabolic or vascular disease requiring statin or other lipid lowering pharmacological or non-pharmacological treatment.
* Total cholesterol > 8, LDL-C > 6 or TG > 6 mmol/L at enrolment

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2007-12; Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Comparison between the active and the placebo group regarding changes in MRI contrast enhancement in terms of the transfer constant (Ktrans) for the carotid region | MRI scan at enrolment visit and within group after 3 months.

SECONDARY OUTCOMES:
Comparison between the active and the placebo group regarding changes in MRI contrast enhancement measured as fractional plasma volume (Vp) and changes in 18FDG uptake in terms of standardised uptake value (SUV), respectively | MRI scan at enrolment visit and within group after 3 months. 18FDG at randomisation visit (baseline) and within group after 3 months treatment.
Change in carotid MRI contrast enhancement in terms of Ktrans and Vp. | At enrolment visit and within group after 3 months treatment.
Change in 18FDG uptake in terms of SUV. | At randomisation visit (baseline) and within group after 3 months treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Håkan Ahlström, MD, Professor, Principal Investigator — Uppsala University Sweden; Maria Leonsson-Zachrissson, MD, Study Physician, Study Chair — AstraZeneca R&D Mölndal
Locations (1):
- Research Site, Uppsala, Sweden